CLINICAL TRIAL: NCT04132089
Title: Incorporating Behavioral Trigger Measures Into a Mobile Health (mHealth) App Design for Chronic Disease Management: Pilot Study in Diabetes
Brief Title: Mobile Health Application for Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Alabama (Other)
Responsible Party: Principal Investigator, Scott Sittig, Assistant Professor, University of South Alabama
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 1122
Record Dates: First submitted 2019-10-08; First posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — capa protein, Drosophila

STUDY DESIGN:
Intervention Model Description: A three factor cross-over design was utilized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): This was the control group for the messaging component of the study (push notifications). These participants only received the mobile health application called capABILITY without messages.
- Facilitator Message Group (Other): This group of participants received the mobile health application called capABILITY and received three facilitator messages per week. Facilitator messages are designed to help people who lack ability to do something.
  Interventions: Behavioral: capABILITY
- Spark Trigger Group (Other): This group of participants received the mobile health application called capABILITY and received three spark messages per week. Spark messages are designed to help people who lack ability to do something.
  Interventions: Behavioral: capABILITY

INTERVENTIONS:
Behavioral: capABILITY — All participants utilized the designed capABILITy application. The application consisted of education material and persuasive messaging. There were two types of messaging components named facilitators and sparks. This created three groups consisting of: control, facilitators and sparks. Participants spent 1 month in each group (total duration of the study was three months).
  Arms: Facilitator Message Group; Spark Trigger Group

SUMMARY:
Creation of a mobile health application for individuals with type II diabetes. This application was designed to improve knowledge, self-efficacy and self-care. The application delivered educational material and provided push notifications (messages). It also allowed for the participants to key in blood glucose levels, carbohydrate consumption and daily exercise.

DETAILED DESCRIPTION:
capABILITY (the mobile health application) was designed to cover three main diabetes content areas which the investigators call modules: diet (module 1), exercise (module 2) and self-management (module 3) (i.e. medication adherence, glucose monitoring). The length of the study was 9 weeks in duration with three weeks of content per module. Within each module new material was delivered each week through capABILITY. Essentially, every Monday started a new week's worth of educational material that was intended to last until Sunday. Each participant was randomly assigned to either the control group (no triggers), spark trigger group or facilitator trigger group. At the beginning of each module the participants would be randomly assigned to one of the three aforementioned classification groups (this was a 2-Factor Cross-Over Design).

The investigators utilized the Perceived Diabetes Self-Efficacy Scale , Diabetes Knowledge Test developed by Michigan University, and the Summary of Diabetes Self-Care Activities Measures scale (SDSCA) . All the participants completed the perceived diabetes self-efficacy scale along with the knowledge test and SDSCA Pre/Post intervention. In addition, the participants answered one self-efficacy, knowledge, self-care and goal question at the conclusion of each week within capABILITY.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 21 years of age or older
* Current diagnosis of type II diabetes
* Must have access to a smartphone and daily internet (WiFi)

Exclusion Criteria:

* Anyone with gestational diabetes

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
20 participants baseline self-efficacy score will be measured at baseline and after the utilization (9 weeks) of the mHealth application capABILITY. | 9 Weeks
  Participants completed the Perceived Diabetes Self-Management Scale at baseline and post intervention to measure their self-efficacy. The measure (scale) consists of eight questions ranging from strongly disagree (1) to strongly agree (5). All items are scored so that high scores equals higher perceived self-efficacy.
20 participants baseline diabetes knowledge score will be measure at baseline and after the utilization (9 weeks) of the mHealth application capABILITY. | 9 Weeks
  Participants completed the Brief Diabetes Knowledge Test (DKT2) at baseline and post intervention to measure their overall type II diabetes knowledge. The measure (scale) consists of twenty- three multiple choice knowledge questions. The score was calculated based on the number of questions answered correctly with higher scores representing a higher knowledge level.
20 participants baseline diabetes self-management score will be measured at baseline and after the utilization (9 weeks) of the mHealth application capABILITY. | 9 Weeks
  Participants completed the Summary of Diabetes Self-Care Activities Questionnaire at baseline and post intervention to measure their diabetes self-care. The measure (scale) consists of twenty five questions ranging from a score of 1 (days per week) to 7 (days per week). All items are scored so that high scores equals higher self-care.

SECONDARY OUTCOMES:
Participants will login and use capABILITY quicker (time measured in seconds) after receiving a behavioral trigger message than those participants who don't receive a behavioral trigger. | 9 Weeks
  Participants will engage quicker with capABILITY after they receive behavioral triggers (Sparks and Facilitators) than those participants who don't receive behavioral triggers. Participants in the Spark and Facilitator groups received push messages (triggers) on Tuesday, Thursday and Saturday at 10:00 am. Time was measured in seconds and the calculation was the time between push notification delivery (10:00am) and the participant login to capABILITY. The smaller the number in seconds the quicker the login time from push notification delivery.
Participants who receive a Spark trigger message will login and use capABILITY quicker (time measured in seconds) than those participants who receive Facilitator trigger message. | 9 Weeks
  Participants will engage quicker with capABILITY after they receive Spark trigger messages than those who receive a Facilitator trigger message. Participants in the Spark and Facilitator groups received push messages (triggers) on Tuesday, Thursday and Saturday at 10:00 am. Time was measured in seconds and the calculation was the time between push notification delivery (10:00am) and the participant login to capABILITY. The smaller the number in seconds the quicker the login time from push notification delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Sittig, PhD, Principal Investigator — University of South Alabama

IPD SHARING:
Plan to Share IPD: No
The participant data from this study will not be shared with other researchers. Findings of the study will be published however.

REFERENCES:
- [Derived] Sittig S, Wang J, Iyengar S, Myneni S, Franklin A. Incorporating Behavioral Trigger Messages Into a Mobile Health App for Chronic Disease Management: Randomized Clinical Feasibility Trial in Diabetes. JMIR Mhealth Uhealth. 2020 Mar 16;8(3):e15927. doi: 10.2196/15927. PMID 32175908